CLINICAL TRIAL: NCT02458742
Title: Spinal Morphine (0.05 mg) Provides an Effective Pain Control in Patients Undergoing Transurethral Resection of Prostate Gland- a Randomized Double-blinded Control Trial
Brief Title: Spinal Morphine Provides an Effective Pain Control in Patients Undergoing Transurethral Resection of Prostate Gland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 019/2558(EC2)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Spinal Anesthesia; Transurethral Resection of Prostate; Analgesia
Keywords: spinal anesthesia; intrathecal morphine; transurethral resection of prostate; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Experimental): 0.5%Bupivacaine 2 ml with morphine 50 mcg for spinal anesthesia
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): 0.5%Bupivacaine 2 ml for spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — 0.5%Hyperbaric bupivacaine 2 ml add morphine 50 mcg for spinal anesthesia
  Other Names: Hyperbaric bupivacaine with morphine
  Arms: Morphine
Drug: Placebo — 0.5%Hyperbaric bupivacaine 2 ml for spinal anesthesia
  Other Names: Hyperbaric bupivacaine
  Arms: Placebo

SUMMARY:
Pain after transurethral resection of prostate is considered mild to moderate severity from detrusor muscle spasm and traction from urinary catheter. Numerous pain relieve methods have been studied including spinal opioids, spinal anesthesia with local anesthetic and dexmedetomidine, periprostatic nerve blockade with bupivacaine and mixing of prilocaine with distilled water irrigation while undergoing a procedure. Most of patients having this procedure are in elderly period, thus many anesthetists avoided spinal morphine which may cause respiratory depressant effect postoperatively. Although previous studies showed effectiveness of spinal morphine 25-200 mcg, some patients suffered from neuraxial opioid side effects.

The aim of this study is to demonstrate efficacy of local anesthetic with intrathecal morphine 50 mcg providing pain relieve after transurethral resection of prostate compare to spinal anesthesia with sole local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Undergoing transurethral resection of prostate gland

Exclusion Criteria:

* Contraindication for spinal anesthesia for any reasons eg. infection, bleeding disorder
* Refuse spinal anesthesia
* Allergic to study drugs
* History of cerebrovascular disease or stroke

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (0-10) | 24 hours postoperatively
  Pain score rating by numerical rating scale in 24-hr postoperative

SECONDARY OUTCOMES:
Requirement of rescue pain | 24 hours postoperatively
  requirement of pain control medication
Adverse effects | 24 hours postoperatively
  incidence of side effects e.g. nausea and vomiting, itching and sedation
Satisfaction score | 24 hours postoperatively
  Satisfaction score rated from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Siriraj Hospital

REFERENCES:
- [Background] Kose O, Saglam HS, Altun ME, Sonbahar T, Kumsar S, Adsan O. Prilocaine irrigation for pain relief after transurethral resection of the prostate. J Endourol. 2013 Jul;27(7):892-5. doi: 10.1089/end.2013.0001. Epub 2013 Jun 12. PMID 23565930
- [Background] Gorur S, Inanoglu K, Akkurt BC, Candan Y, Kiper AN. Periprostatic nerve blockage reduces postoperative analgesic consumption and pain scores of patients undergoing transurethral prostate resection. Urol Int. 2007;79(4):297-301. doi: 10.1159/000109712. PMID 18025845
- [Background] Kim JE, Kim NY, Lee HS, Kil HK. Effects of intrathecal dexmedetomidine on low-dose bupivacaine spinal anesthesia in elderly patients undergoing transurethral prostatectomy. Biol Pharm Bull. 2013;36(6):959-65. doi: 10.1248/bpb.b12-01067. PMID 23727917
- [Background] Suksompong S, Pongpayuha P, Lertpaitoonpan W, von Bormann B, Phanchaipetch T, Sanansilp V. Low-dose spinal morphine for post-thoracotomy pain: a prospective randomized study. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):417-22. doi: 10.1053/j.jvca.2012.12.003. Epub 2013 Mar 29. PMID 23545346
- [Background] Duman A, Apiliogullari S, Balasar M, Gurbuz R, Karcioglu M. Comparison of 50 microg and 25 microg doses of intrathecal morphine on postoperative analgesic requirements in patients undergoing transurethral resection of the prostate with intrathecal anesthesia. J Clin Anesth. 2010 Aug;22(5):329-33. doi: 10.1016/j.jclinane.2009.09.006. PMID 20650378
- [Background] Kirson LE, Goldman JM, Slover RB. Low-dose intrathecal morphine for postoperative pain control in patients undergoing transurethral resection of the prostate. Anesthesiology. 1989 Aug;71(2):192-5. doi: 10.1097/00000542-198908000-00004. PMID 2667399
- [Background] Ozbek H, Deniz MN, Erakgun A, Erhan E. Comparison of 75 and 150 mug doses of intrathecal morphine for postoperative analgesia after transurethral resection of the prostate under spinal anesthesia. J Opioid Manag. 2013 Nov-Dec;9(6):415-20. doi: 10.5055/jom.2013.0184. PMID 24481930
- [Background] Sakai T, Use T, Shimamoto H, Fukano T, Sumikawa K. Mini-dose (0.05 mg) intrathecal morphine provides effective analgesia after transurethral resection of the prostate. Can J Anaesth. 2003 Dec;50(10):1027-30. doi: 10.1007/BF03018367. PMID 14656781